CLINICAL TRIAL: NCT02466646
Title: Evaluation of Gingival Crevicular Fluid Interleukin-1β and Interleukin-17 Levels and Periodontal Pathogens After Full-Mouth Disinfection Initial Periodontal Treatment in Generalized Aggressive Periodontitis Patients
Brief Title: Evaluation of Efficacy of Full-mouth Disinfection in Generalized Aggressive Periodontitis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAG-C-DRP-280214-0043
Record Dates: First submitted 2015-05-27; First posted 2015-06-09 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Aggressive Periodontitis
Keywords: Periodontal Debridement; Gingival Crevicular Fluid; Aggressive Periodontitis; Interleukin-1beta; Interleukin-17; Bacteria
MeSH Terms: conditions — Aggressive Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Full-mouth Disinfection IPT (Active Comparator): Initial periodontal treatment was performed in 2 sessions with application of chlorhexidine to the intra-oral niches within 24 hours (Klorhex® Gel 1% for 10 minutes, Klorhex® Spray 0,2% and Klorhex® rinse 0,2% for 3 weeks).
  Interventions: Drug: Klorhex® Gel, rinse and spray
- Conventional IPT (Experimental): Initial periodontal treatment was performed in a quadrant-wise manner at 1-week intervals.
  Interventions: Procedure: Conventional IPT
- Full-mouth IPT (Experimental): Initial periodontal treatment was performed in 2 sessions within 24 hours.
  Interventions: Procedure: Full-mouth IPT

INTERVENTIONS:
Drug: Klorhex® Gel, rinse and spray — Initial periodontal treatment was performed in 2 sessions with application of chlorhexidine to the intra-oral niches within 24 hours (Klorhex® Gel 1% for 10 minutes, Klorhex® Spray 0,2% and Klorhex® rinse 0,2% for 3 weeks).
  Other Names: FMD
  Arms: Full-mouth Disinfection IPT
Procedure: Conventional IPT — Initial periodontal treatment was performed in a quadrant-wise manner at 1-week intervals.
  Other Names: Q-SRP
  Arms: Conventional IPT
Procedure: Full-mouth IPT — Initial periodontal treatment was performed in 2 sessions within 24 hours.
  Other Names: FM-SRP
  Arms: Full-mouth IPT

SUMMARY:
The purpose of this study is to determine whether full-mouth disinfection is effective in the initial periodontal treatment of generalized aggressive periodontitis on clinical parameters, gingival crevicular fluid interleukin-1β (IL-1β) and interleukin-17 (IL-17) and periodontal pathogen levels compared with conventional initial periodontal treatment and full-mouth initial periodontal treatment.

The investigators' hypothesis is to test whether full-mouth disinfection in the initial periodontal treatment of generalized aggressive periodontitis enhance the clinical, biochemical and microbiological parameters in comparison to conventional initial periodontal treatment and full-mouth initial periodontal treatment.

DETAILED DESCRIPTION:
The present study aimed to compare the efficacy of conventional initial periodontal treatment (C-IPT), full-mouth disinfection IPT (FMD-IPT) and full-mouth IPT (FM-IPT) and the levels of gingival crevicular fluid interleukin-1β (IL-1β) and interleukin-17 (IL-17), Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Fusobacterium nucleatum, Prevotella intermedia, Parvimonas micra and Campylobacter rectus in patients with generalized aggressive periodontitis (GAgP) over 6-months period. Forty-two GAgP patients were randomly assigned into 3 groups. IPT was performed in a quadrant-wise manner at 1-week intervals in C-IPT, in 2 sessions within 24 hours in FM-IPT, and in 2 sessions with application of chlorhexidine to the intra-oral niches within 24 hours in FMD-IPT. FMD-IPT group also used daily 0,2% chlorhexidine for 3 weeks. At baseline, 3 and 6 months clinical parameters consisting of plaque index, gingival index, probing depth, bleeding on probing and clinical attachment level were recorded, gingival crevicular fluid and microbiological samples were collected. Gingival crevicular fluid levels of IL-1β and IL-17 were analyzed using ELISA. The quantitative real-time polymerase chain reaction method was used for the quantitative detection of periodontal pathogens.

ELIGIBILITY:
Inclusion Criteria:

* No systemic diseases that could influence the outcome of the therapy
* No smoking
* No medications affecting periodontal tissues
* No pregnancy or lactation
* Presence of at least 15 teeth

Exclusion Criteria:

* Received antibiotic treatment in the previous 3 months
* Smokers
* Pregnancy and lactation
* Received periodontal treatment in the previous 6 months
* Presence of less than 15 teeth
* Presence of systemic diseases

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2012-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Basak Dogan, Prof. Dr., Study Director — Marmara University, Faculty of Dentistry, Department of Periodontology; Dilek Mamaklioglu, Dr., Principal Investigator — Marmara University, Faculty of Dentistry, Department of Periodontology

REFERENCES:
- [Background] Aimetti M, Romano F, Guzzi N, Carnevale G. Full-mouth disinfection and systemic antimicrobial therapy in generalized aggressive periodontitis: a randomized, placebo-controlled trial. J Clin Periodontol. 2012 Mar;39(3):284-94. doi: 10.1111/j.1600-051X.2011.01795.x. Epub 2012 Jan 4. PMID 22220822
- [Background] Mongardini C, van Steenberghe D, Dekeyser C, Quirynen M. One stage full- versus partial-mouth disinfection in the treatment of chronic adult or generalized early-onset periodontitis. I. Long-term clinical observations. J Periodontol. 1999 Jun;70(6):632-45. doi: 10.1902/jop.1999.70.6.632. PMID 10397519
- [Background] de Lima Oliveira AP, de Faveri M, Gursky LC, Mestnik MJ, Feres M, Haffajee AD, Socransky SS, Teles RP. Effects of periodontal therapy on GCF cytokines in generalized aggressive periodontitis subjects. J Clin Periodontol. 2012 Mar;39(3):295-302. doi: 10.1111/j.1600-051X.2011.01817.x. Epub 2011 Nov 30. PMID 22126282

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total of 54 subjects were assessed for eligibility. Prior to assignment of participants, 2 subjects declined to participate and 10 participants were not meeting inclusion criteria
Groups:
- Full-mouth Disinfection IPT: Initial periodontal treatment was performed in 2 sessions with application of chlorhexidine to the intra-oral niches within 24 hours (Klorhex® Gel 1% for 10 minutes, Klorhex® Sprey 0,2% and Klorhex® rinse 0,2% for 3 weeks).
Period: Overall Study
Arm/Group | Full-mouth Disinfection IPT | Conventional IPT | Full-mouth IPT
Started | 14 | 14 | 14
Completed | 14 | 14 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Full-mouth Disinfection IPT | Conventional IPT | Full-mouth IPT | Total
Number analyzed (Participants) | 14 | 14 | 14 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.64 (5.65) | 29.86 (6.41) | 31.86 (4.56) | 29.45 (5.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 8 | 25
  Male | 4 | 7 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 14 | 14 | 14 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 14 | 14 | 14 | 42
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Probing Depth
Time Frame: 6 months after initial periodontal treatment
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Full-mouth Disinfection IPT | Conventional IPT | Full-mouth IPT
Number analyzed (Participants) | 14 | 14 | 14
mm
  Baseline Probing Depth (PD) | 4.55 (0.72) | 4.80 (0.62) | 4.90 (0.62)
  6th month PD | 2.71 (0.29) | 3.40 (0.50) | 3.04 (0.39)
Statistical Analysis 1: Comparison: Full-mouth Disinfection IPT vs Conventional IPT vs Full-mouth IPT; Test type: Other; p < 0.01, Kruskal-Wallis — The threshold for statistical significance was p=0.05; Mean Difference (Net) = 0.30

2. Secondary Outcome: Gingival Crevicular Fluid Interleukin-1β and Interleukin-17 Levels (pg)
Time Frame: Baseline, 3 and 6 months after initial periodontal treatment
Measure: Mean (Standard Deviation); unit: Picogram
Arm/Group | Full-mouth Disinfection IPT | Conventional IPT | Full-mouth IPT
Number analyzed (Participants) | 14 | 14 | 14
Picogram
  Baseline Interleukin-1β | 2.53 (0.39) | 2.27 (0.62) | 2.15 (0.64)
  3rd month IL-1β | 2.07 (0.51) | 2.11 (0.39) | 2.06 (0.24)
  6th month IL-1β | 2.11 (0.55) | 1.90 (0.49) | 1.96 (0.47)
  Baseline Interleukin-17 | 18.53 (7.29) | 19.91 (10.68) | 19.67 (7.60)
  3rd month IL-17 | 21.07 (10.94) | 21.02 (9.94) | 19.76 (4.83)
  6th month IL-17 | 20.05 (7.49) | 19.27 (7.56) | 18.46 (4.61)
Statistical Analysis 1: Comparison: Full-mouth Disinfection IPT vs Conventional IPT vs Full-mouth IPT; Test type: Other; p > 0.05, Kruskal-Wallis — The threshold for statistical significance was P=0.05; Mean Difference (Net) = 2

3. Secondary Outcome: Level of A. Actinomycetemcomitans
Time Frame: Baseline, 3 and 6 months after initial periodontal treatment
Measure: Mean (Standard Deviation); unit: log10(cells/ml)
Arm/Group | Full-mouth Disinfection IPT | Conventional IPT | Full-mouth IPT
Number analyzed (Participants) | 14 | 14 | 14
log10(cells/ml)
  Baseline A. actinomycetemcomitans level | 3.65 (1.21) | 3.84 (1.20) | 3.63 (1.26)
  3rd months A. actinomycetemcomitans level | 3.27 (0.71) | 3.73 (1.28) | 3.47 (1.10)
  6th month A. actinomycetemcomitans level | 2.92 (0.64) | 3.59 (1.10) | 3.47 (1.21)
Statistical Analysis 1: Comparison: Full-mouth Disinfection IPT vs Conventional IPT vs Full-mouth IPT; Test type: Other; p = 0.229, Kruskal-Wallis — Threshold for statistical significance is p=0.05

4. Secondary Outcome: Level of Porphyromonas Gingivalis
Time Frame: Baseline, 3 and 6 months after initial periodontal treatment
Measure: Mean (Standard Deviation); unit: log10(cells/ml)
Arm/Group | Full-mouth Disinfection IPT | Conventional IPT | Full-mouth IPT
Number analyzed (Participants) | 14 | 14 | 14
log10(cells/ml)
  Baseline P. gingivalis level | 4.64 (1.47) | 5.50 (0.71) | 5.47 (1.06)
  3rd months P. gingivalis level | 2.90 (0.50) | 3.60 (1.15) | 3.74 (1.05)
  6th month P. gingivalis level | 3.25 (0.98) | 4.00 (1.13) | 3.84 (0.76)
Statistical Analysis 1: Comparison: Full-mouth Disinfection IPT vs Conventional IPT vs Full-mouth IPT; Test type: Other; p = 0.280, Kruskal-Wallis — Threshold for statistical significance is p=0.05

5. Secondary Outcome: Level of Fusobacterium Nucleatum
Time Frame: Baseline, 3 and 6 months after initial periodontal treatment
Measure: Mean (Standard Deviation); unit: log10(cells/ml)
Arm/Group | Full-mouth Disinfection IPT | Conventional IPT | Full-mouth IPT
Number analyzed (Participants) | 14 | 14 | 14
log10(cells/ml)
  Baseline F. nucleatum level | 4.67 (0.66) | 4.78 (0.45) | 4.66 (0.51)
  3rd month F. nucleatum level | 3.84 (0.55) | 3.99 (0.76) | 4.42 (0.68)
  6th month F. nucleatum level | 3.73 (1.00) | 3.84 (1.03) | 4.17 (0.61)
Statistical Analysis 1: Comparison: Full-mouth Disinfection IPT vs Conventional IPT vs Full-mouth IPT; Test type: Other; p = 0.712, Kruskal-Wallis; Threshold for statistical significance is p=0.05

6. Secondary Outcome: Level of Parvimonas Micra
Time Frame: Baseline, 3 and 6 months after initial periodontal treatment
Measure: Mean (Standard Deviation); unit: log10(cells/ml)
Arm/Group | Full-mouth Disinfection IPT | Conventional IPT | Full-mouth IPT
Number analyzed (Participants) | 14 | 14 | 14
log10(cells/ml)
  Baseline P. micra level | 4.96 (0.50) | 4.86 (0.45) | 4.70 (0.58)
  3rd month P. micra level | 4.22 (0.49) | 4.34 (0.43) | 4.51 (0.52)
  6th month P. micra level | 4.28 (0.63) | 4.30 (0.58) | 4.43 (0.70)
Statistical Analysis 1: Comparison: Full-mouth Disinfection IPT vs Conventional IPT vs Full-mouth IPT; Test type: Other; p = 0.674, Kruskal-Wallis — The threshold for statistical significance is p=0.05

7. Secondary Outcome: Bleeding on Probing
Description: Possible score for BOP range from %0 (no sites with bleeding on probing) to %100 (all sites with bleeding on probing). Higher scores mean worse outcome.
Time Frame: Baseline, 3 and 6 months after initial periodontal treatment
Measure: Mean (Standard Deviation); unit: percentage of BOP positive sites
Arm/Group | Full-mouth Disinfection IPT | Conventional IPT | Full-mouth IPT
Number analyzed (Participants) | 14 | 14 | 14
percentage of BOP positive sites
  Baseline Bleeding on Probing (BOP) | 78.30 (15.05) | 89.28 (9.03) | 85.77 (13.49)
  3rd month BOP | 38.87 (7.15) | 54.43 (14.80) | 48.90 (10.47)
  6th month BOP | 42.78 (5.91) | 60.19 (16.33) | 49.74 (13.03)
Statistical Analysis 1: Comparison: Full-mouth Disinfection IPT vs Conventional IPT vs Full-mouth IPT; Test type: Other; p = 0.006, Kruskal-Wallis — The threshold for statistical significance was p=0.05; Mean Difference (Net) = 30

8. Secondary Outcome: Plaque Index
Description: Possible scores for Plaque Index range from 0 (no plaque) to 3 (visible plaque all around the tooth). Higher scores mean a worse outcome
Time Frame: Baseline, 3 and 6 months after initial periodontal treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Full-mouth Disinfection IPT | Conventional IPT | Full-mouth IPT
Number analyzed (Participants) | 14 | 14 | 14
score on a scale
  Baseline PI | 1.51 (0.28) | 1.76 (0.31) | 1.62 (0.20)
  3rd month PI | 0.67 (0.12) | 0.69 (0.18) | 0.84 (0.13)
  6th month PI | 0.72 (0.16) | 0.77 (0.20) | 0.82 (0.20)
Statistical Analysis 1: Comparison: Full-mouth Disinfection IPT vs Conventional IPT vs Full-mouth IPT; Test type: Other; p = 0.373, Kruskal-Wallis; Mean Difference (Net) = 0.5

9. Secondary Outcome: Gingival Index
Description: Possible score for Gingival Index range from 0 (healthy gingiva) to 3 (severe gingivitis with bleeding). Higher scores mean worse outcome
Time Frame: Baseline, 3 and 6 months after initial periodontal treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Full-mouth Disinfection IPT | Conventional IPT | Full-mouth IPT
Number analyzed (Participants) | 14 | 14 | 14
score on a scale
  Baseline GI | 1.61 (0.28) | 1.80 (0.22) | 1.74 (0.23)
  3rd month GI | 1.17 (0.10) | 1.15 (0.29) | 1.24 (0.09)
  6th month GI | 1.20 (0.06) | 1.29 (0.21) | 1.21 (0.10)
Statistical Analysis 1: Comparison: Full-mouth Disinfection IPT vs Conventional IPT vs Full-mouth IPT; Test type: Other; p = 0.528, Kruskal-Wallis; Mean Difference (Net) = 0.6

10. Secondary Outcome: Clinical Attachment Level
Time Frame: Baseline, 3 and 6 months after initial periodontal treatment
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Full-mouth Disinfection IPT | Conventional IPT | Full-mouth IPT
Number analyzed (Participants) | 14 | 14 | 14
mm
  Baseline Clinical Attachment Level (CAL) | 5.20 (0.93) | 5.67 (1.24) | 5.79 (0.67)
  3rd month CAL | 4.54 (0.75) | 4.94 (1.24) | 5.10 (0.75)
  6th month CAL | 4.51 (0.69) | 5.25 (1.37) | 5.13 (0.77)
Statistical Analysis 1: Comparison: Full-mouth Disinfection IPT vs Conventional IPT vs Full-mouth IPT; Test type: Other; p = 0.208, Kruskal-Wallis; Mean Difference (Net) = 1

11. Secondary Outcome: Level of Prevotella Intermedia
Time Frame: Baseline, 3 and 6 months after initial periodontal treatment
Measure: Mean (Standard Deviation); unit: log10(cells/ml)
Arm/Group | Full-mouth Disinfection IPT | Conventional IPT | Full-mouth IPT
Number analyzed (Participants) | 14 | 14 | 14
log10(cells/ml)
  Baseline P. intermedia level | 4.24 (1.07) | 5.51 (0.86) | 4.84 (0.98)
  3rd month P. intermedia level | 2.73 (0.79) | 3.70 (1.20) | 3.81 (1.40)
  6th month P. intermedia level | 2.98 (0.75) | 4.14 (1.19) | 3.46 (0.97)
Statistical Analysis 1: Comparison: Full-mouth Disinfection IPT vs Conventional IPT vs Full-mouth IPT; Test type: Other; p = 0.051, Kruskal-Wallis

12. Secondary Outcome: Level of Campylobacter Rectus
Time Frame: Baseline, 3 and 6 months after initial periodontal treatment
Measure: Mean (Standard Deviation); unit: log10(cells/ml)
Arm/Group | Full-mouth Disinfection IPT | Conventional IPT | Full-mouth IPT
Number analyzed (Participants) | 14 | 14 | 14
log10(cells/ml)
  Baseline C. rectus level | 5.95 (0.70) | 6.19 (0.60) | 5.99 (0.72)
  3rd month C. rectus level | 4.63 (0.79) | 5.01 (1.04) | 5.25 (0.87)
  6th month C. rectus level | 4.64 (0.82) | 4.99 (1.15) | 5.03 (0.93)
Statistical Analysis 1: Comparison: Full-mouth Disinfection IPT vs Conventional IPT vs Full-mouth IPT; Test type: Other; p = 0.647, Kruskal-Wallis — The threshold for statistical significance is p=0.05

ADVERSE EVENTS:
Time Frame: 6 months
Description: Only Other (Not Including Serious) Adverse Events were monitored, Serious Adverse Events were not monitored.
Arm/Group | Full-mouth Disinfection IPT | Conventional IPT | Full-mouth IPT
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No